CLINICAL TRIAL: NCT05430347
Title: A Multicenter Phase II Clinical Study of Pyrotinib or Pertuzumab Combined With Docetaxel, Carboplatin, and Trastuzumab in Neoadjuvant Therapy for HR-positive, HER2-positive Breast Cancer
Brief Title: Clinical Study of Pyrotinib in Neoadjuvant Therapy of HR-positive and HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pyrotinib neoadjuvant
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: HR+/HER2+ Breast cancer; Neoadjuvant therapy; pyrotinib
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The treatment regimen of the experimental group was pyrotinib combined with docetaxel, carboplatin and trastuzumab, while the treatment regimen of the control group was pertuzumab combined with docetaxel, carboplatin and trastuzumab (the control group was standard treatment). Surgical treatment was performed after 6 courses of neoadjuvant therapy
Masking Description: This study is an open-design, multicenter, randomized controlled prospective clinical study with 80 patients. Subjects will be randomly assigned 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCbHPy*6 (Experimental): Pyrotinib combined with docetaxel, carboplatin and trastuzumab for 6 cycles (Every three weeks).
  T (Docetaxel 100 mg/m2, d1) C (Carboplatin, AUC 6, D1) H (Trastuzumab, 8 mg/kg for the first dose, 6 mg/kg for the rest, D1) Py (pyrotinib 400mg, qD, D1-21)
  Interventions: Combination Product: Neoadjuvant therapy: TCbHPy
- TCbHP*6 (Active Comparator): Pertuzumab combined with docetaxel, carboplatin and trastuzumab for 6 cycles (Every three weeks).
  T (Docetaxel 100 mg/m2, d1) C (Carboplatin, AUC 6, D1) H (Trastuzumab, 8 mg/kg for the first dose, 6 mg/kg for the rest, D1) P (Pertuzumab, 840mg for the first dose, 420mg for the rest, D1))
  Interventions: Combination Product: Neoadjuvant therapy: TCbHP

INTERVENTIONS:
Combination Product: Neoadjuvant therapy: TCbHPy — Pyrotinib combined with docetaxel, carboplatin and trastuzumab (TCbHPy) for neoadjuvant therapy of HR+/HER2+ breast cancer
  Arms: TCbHPy*6
Combination Product: Neoadjuvant therapy: TCbHP — Pertuzumab combined with docetaxel, carboplatin and trastuzumab (TCbHP) for neoadjuvant therapy of HR+/HER2+ breast cancer
  Arms: TCbHP*6

SUMMARY:
Due to neoadjuvant therapy with trastuzumab and pertuzumab is less effective for HR+/HER2+ breast cancer, and the PHEDRA Clinical Study subgroup analysis showed that the addition of pyrotinib to trastuzumab more than doubled pCR rates in HR+/HER2+ patients. our research group proposed a hypothesis that pyrotinib may be more advantageous for HR+/HER2+ breast cancer. Therefore, our center intends to carry out a multi-center, randomized controlled, prospective clinical study to compare the efficacy of pyrotinib or pertuzumab combined with docetaxel, carboplatin and trastuzumab in neoadjuvant therapy for patients with HR+/HER2+ breast cancer, and to conduct a comparative study on the safety.

DETAILED DESCRIPTION:
Different anti-HER2-targeting drugs act on different parts and types of HER2 molecules, so their mechanisms and effects are different. Trastuzumab and pertuzumab are the most commonly used anti-HER2 targeting drugs, which target the extracellular segment of THE HER2 molecule. The major guidelines recommend the use of trastuzumab and pertuzumab in the use of neoadjuvant therapy with a two-target regimen. Another commonly used class of anti-HER2-targeting drugs are Tyrosine kinase inhibitors (TKI), which target the intracellular segment of the HER2 molecule. Not only that, take domestically developed pyrotinib as an example, in addition to targeting HER2, it also targets HER1 and HER4. Because of the different mechanisms of action, TKI is still effective in patients with trastuzumab and/or pertuzumab resistant relapsing metastasis. To investigate the efficacy of pyrotinib in neoadjuvant therapy, a prospective, randomized, double-blind, multicenter clinical trial, the PHEDRA Clinical Study, was conducted in China. Results presented at the 2021 ASCO Meeting showed that addition of pyrotinib to trastuzumab also significantly increased tpCR rate (22.0% vs 41.0%; P < 0.0001), and the pCR rate was similar to trastuzumab + pertuzumab double target (39.3% for Neosphere and Peony). Based on these results, neoadjuvant therapy regimens with trastuzumab and TKI have been included in the 2022 CSCO guidelines.

Of note, there were also differences in Hormone Receptor (HR) status in patients with HER2-positive breast cancer. After neoadjuvant chemotherapy combined with trastuzumab and pertuzumab double-target therapy, the pCR rate of HR-/HER2+ breast cancer was higher than HR+/HER2+ breast cancer. In contrast, a PHEDRA subgroup analysis showed that the addition of pyrotinib to trastuzumab more than doubled pCR rates in HR+/HER2+ patients (29.9% vs 12.2%) . In addition, in another adjunctive study of TKI drug neratinib, subgroup results also suggested that neratinib had a better effect on HR+/HER2+.

Based on the above results, our research group proposed a hypothesis that TKI drugs may be more advantageous for HR+/HER2+ breast cancer. Therefore, our center intends to carry out a multi-center, randomized controlled, prospective clinical study to compare the efficacy of pyrotinib or pertuzumab combined with docetaxel, carboplatin and trastuzumab in neoadjuvant therapy for patients with HR+/HER2+ breast cancer, and to conduct a comparative study on the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 with breast cancer;
2. Pathologically confirmed unilateral invasive ductal carcinoma (with or without intraductal carcinoma components);
3. Proposed to receive neoadjuvant therapy;
4. Positive ER and/or PgR (defined as ≥10% positive immunohistochemical test);
5. HER2 positive (defined as IMMUNOHISTOchemical HER2 ++, or HER2 ++ and in situ hybridization (ISH) results in HER2 gene amplification);
6. There is no evidence of metastasis in clinical or imaging;
7. ECOG score 0 or 1;
8. White blood cell count ≥3.5×109/L, neutrophil count ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥90 g/L before neoadjuvant therapy;
9. Before neoadjuvant therapy, AST and ALT < 1.5 times the upper limit of normal value, alkaline phosphatase < 2.5 times the upper limit of normal value, total bilirubin < 1.5 times the upper limit of normal value; Serum creatinine < 1.5 times the upper limit of normal value;
10. LVEF≥55% on 2d echocardiography before neoadjuvant therapy;
11. Signed informed consent.

Exclusion Criteria:

1. Clinical or imaging suspicion of lateral breast malignancy has not been confirmed;
2. Prior malignancy (except basal cell carcinoma of the skin and carcinoma in situ of the cervix), including contralateral breast cancer;
3. The patient has been enrolled in other clinical trials;
4. Patients suffering from serious systemic diseases and/or uncontrollable infections cannot be enrolled in the study;
5. Severe cardiovascular and cerebrovascular diseases (e.g., unstable angina pectoris, chronic heart failure, uncontrolled hypertension > 150/90mmHg, myocardial infarction or cerebrovascular accident) within the first 6 months of randomization;
6. Have a history of blood system diseases, especially platelet-related diseases;
7. Patients with previous intestinal inflammation, intestinal dysfunction, severe diarrhea and constipation;
8. People who are known to be allergic to chemotherapy drugs, targeted drugs or TKI drugs;
9. Women of childbearing age refuse contraception during treatment and within 8 weeks after completion of treatment;
10. Pregnant and lactation women;
11. positive pregnancy test before drug use after joining the test;
12. Mental illness, cognitive impairment, inability to understand the test protocol and side effects, inability to complete the test protocol and follow-up workers (systematic evaluation is required before the trial is enrolled);
13. Persons without personal freedom and independent capacity for civil conduct.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
tpCR rate (ypT0/is ypN0) | 1 month after surgery
  Pathological complete response rate after neoadjuvant ( both breast and axillary lymph nodes, in which the breast may have residual carcinoma in situ)

SECONDARY OUTCOMES:
iDFS | 3 years
  invasive Disease Free Survival
EFS | 3 years
  Event Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No